CLINICAL TRIAL: NCT03265171
Title: A Single-patient Study of Repeat-dose Administration of ProMetic Plasminogen (Human) Intravenous Infusion in an Adult With Hypoplasminogenemia
Brief Title: A Single-patient Study of Repeat-dose Administration of Prometic Plasminogen (Human) Intravenous
Status: No longer available | Type: Expanded Access
Sponsor: Prometic Biotherapeutics, Inc. (Industry)
Collaborators: Cedars-Sinai Medical Center (Other); Vanderbilt University Medical Center (Other); Indiana Hemophilia &Thrombosis Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2002C013G
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hypoplasminogenemia
MeSH Terms: conditions — Congenital Plasminogen Deficiency | interventions — Plasminogen

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Plasminogen (Human)

SUMMARY:
These are single-patient studies with repeat-dose administration of ProMetic Plasminogen IV infusion in one adult and one child with hypoplasminogenemia. These patients are under treatment to address wound healing and obstructions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided informed consent.
* Patient has a diagnosis of compound homozygous Type 1 plasminogen deficiency as evidence by ligneous conjunctivitis since birth as well as involvement of the conjunctiva, nasopharynx, gingiva, tracheobronchial tree, gastrointestinal tract, and urinary tract.

Exclusion Criteria:

* Not applicable

Min Age: 16 Months | Sex: All
Age Groups: Child, Adult, Older Adult